CLINICAL TRIAL: NCT02710851
Title: A PhaseⅡ Randomized, Double-Blinded, Placebo Controlled Study to Evaluate the Immunogenicity of the Recombinant (E.Coli) Human Papillomavirus Type 6/11 Bivalent Vaccine in Healthy Volunteers Aged 18-55 Years
Brief Title: Immunogenicity Study of the Recombinant Human Papillomavirus Virus Type 6/11 Bivalent Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPV-PRO-005
Record Dates: First submitted 2016-01-27; First posted 2016-03-17 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Condylomata Acuminata
Keywords: human papillomavirus vaccine; condylomata acuminata
MeSH Terms: conditions — Condylomata Acuminata | interventions — hecolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- low dosage HPV Vaccine(1:1) (Experimental): Participants in this arm would receive low dosage HPV vaccine with virus-like particles type 6 and 11 at 1:1 ratio.
  Interventions: Biological: low dosage HPV Vaccine(1:1)
- low dosage HPV Vaccine(1:2) (Experimental): Participants in this arm would receive low dosage HPV vaccine with virus-like particles type 6 and 11 at 1:2 ratio.
  Interventions: Biological: low dosage HPV Vaccine(1:2)
- high dosage HPV Vaccine(1:1) (Experimental): Participants in this arm would receive high dosage HPV vaccine with virus-like particles type 6 and 11 at 1:1 ratio.
  Interventions: Biological: high dosage HPV Vaccine(1:1)
- Hepatitis E vaccine,Hecolin® (Placebo Comparator): Participants in this arm would receive Hepatitis E vaccine,Hecolin®
  Interventions: Biological: Hepatitis E vaccine,Hecolin®

INTERVENTIONS:
Biological: low dosage HPV Vaccine(1:1) — Participants would intramuscularly receive low dosage HPV bivalent vaccine with virus-like particles type 6 and 11 at 1:1 ratio.
  All participants would be invited to receive 3 doses vaccine at 0, 1, 6 month.
  Arms: low dosage HPV Vaccine(1:1)
Biological: low dosage HPV Vaccine(1:2) — Participants would intramuscularly receive low dosage HPV bivalent vaccine with virus-like particles type 6 and 11 at 1:2 ratio.
  All participants would be invited to receive 3 doses vaccine at 0, 1, 6 month.
  Arms: low dosage HPV Vaccine(1:2)
Biological: high dosage HPV Vaccine(1:1) — Participants would intramuscularly receive high dosage HPV bivalent vaccine with virus-like particles type 6 and 11 at 1:1 ratio.
  All participants would be invited to receive 3 doses vaccine at 0, 1, 6 month.
  Arms: high dosage HPV Vaccine(1:1)
Biological: Hepatitis E vaccine,Hecolin® — Participants would intramuscularly receive Hepatitis E vaccine for 3 doses at 0, 1, 6 month.
  Arms: Hepatitis E vaccine,Hecolin®

SUMMARY:
This phase Ⅱ clinical study was designed to evaluate the immunogenicity and safety of the novel recombinant HPV type 6/11 bivalent vaccine, manufactured by Xiamen Innovax Biotech CO., LTD., in healthy volunteers aged 18-55 years of age at enrollment. The study volunteers would be randomized to receive the 3 different formulations of the novel HPV vaccine or placebo vaccine (recombinant hepatitis E vaccine) administered intramuscularly according to a 0-1-6 month schedule. This is a double-blind study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged between 18 and 55 years.
2. Judged as healthy and eligible for vaccination by the investigators through a self-reported medical history and some physical examinations.
3. Written informed consent obtained from the participants.
4. Able to comply with the requests of the study.
5. Axillary temperature not higher than 37.0°C
6. Non-pregnancy verified by a urine pregnancy test.

Exclusion Criteria:

1. Pregnant or breastfeeding or plan to be pregnant within 7 months.
2. Use of any investigational product or non-registered product (drug or vaccine) within 30 days preceding the first dose of the study vaccine or plan to use during the study period.
3. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment.
4. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine.
5. Administration of any attenuated live vaccines within 30 days preceding the first dose of the study vaccine or any subunit or inactivated vaccines within 14 days before vaccination.
6. Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination.
7. Having the plan to participate another clinical trial during the study period.
8. Received another HPV vaccine.
9. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, .or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response).
10. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy, urticaria, dyspnea, angioneurotic edema or abdominal pain.
11. Having serious disease of internal medicine, such as hypertension, cardiac disease, diabetes, hyperthyroidism et al.
12. Asthma that required emergent treatment, hospitalization, oral or intravenous corticosteroid for unstable condition within the past 2 years.
13. Diagnosed coagulant function abnormality (i.e., clotting factors absent, clotting hemorrhagic disease, abnormal platelet function) or blood coagulation disorder.
14. Epilepsy, except fever epilepsy at under 2 years of age, alcohol-induced epilepsy in 3 years before abstinence, or idiopathic epilepsy requiring no treatment in the past 3 years.
15. Past or current two-stage affective psychosis, not well controlled in the past 2 years or requiring drugs, or h a tendency to commit suicide.
16. Other medical, psychological, social or occupational factors that, according to the investigators' judgment, might affect the individual's ability to obey the protocol or sign the informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 640 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Anti-HPV 6 and anti-HPV 11 seroconversion rates (type specific IgG antibody) | 7 months
Anti-HPV 6 and anti-HPV 11 geometric mean concentrations (type specific IgG antibody) | 7 months

SECONDARY OUTCOMES:
Number of serious adverse events throughout the study | 7 months
  All the serious adverse events throughout the study would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Master, Study Chair — Xiamen University; Yuemei Hu, Bachelor, Principal Investigator — Jiangsu center for Disease Prevention and Control